CLINICAL TRIAL: NCT04121949
Title: A Prospective, Randomized, Controlled, Parallel-group, Multicentre Trial to Examine the Cost-effectiveness and Safety of Adding the CADScorSystem as a Rule-out Test in Patients Referred With Symptoms Suggestive of Stable Coronary Artery Disease.
Brief Title: Cost-effectiveness and Safety of the CADScorSystem in Patients With Symptoms Suggestive of Stable Coronary Artery Disease.
Acronym: FILTER-SCAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Region Hovedstadens Apotek (Other Government); Larix A/S (Industry); Acarix (Industry); Kai Hansen Foundation (Other); Kai Houmann Nielsens Fond (Other)
Responsible Party: Principal Investigator, Eva Prescott, Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FILTER-SCAD
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Angina, Stable
Keywords: coronary artery disease; diagnostic strategies
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, controlled, multicentre, superiority trial with two parallel groups including patients with symptoms suggestive of stable CAD at a low-to-intermediate likelihood of obstructive CAD (pre-test probability of 0-85%). Subjects will be randomized 1:1 to either (1) standard diagnostic strategy according to current guidelines, i.e. DF-score stratification followed by NIT, if indicated, or (2) DF-score plus CAD-score stratification followed by NIT, if indicated.
Who Masked: Outcomes Assessor
Masking Description: Allocation will be hidden from the independent Clinical Events Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive standard-of-care treatment recommended by current ESC guidelines for patients with low to intermediate likelihood of stable CAD using the Diamond-Forrester (DF) score only: Rule-out if DF-score <15%; NIT if DF-score 15-85%.
  As per January 2020 the protocol was updated according to the 2019 ESC Guidelines on Chronic Coronary Syndrome:
  The control group will receive standard-of-care treatment recommended by current ESC guidelines based on the patients likelihood of stable CAD using the Pre-test Probability score (PTP): Rule-out if PTP≤5%, NIT may be considered if PTP 6-15%, NIT if PTP>15%
- Intervention group (Experimental): The intervention group will undergo a modified diagnostic pathway where a CAD-score <30 rules out stable CAD in the group of patients having a DF-score <15% and a CAD-score ≤20 rules out stable CAD in the group of patients having a DF-score in the range 15-85%, and thus not tested with NIT. Otherwise NIT is performed.
  As per January 2020 the protocol was updated according to the 2019 ESC Guidelines on Chronic Coronary Syndrome:
  The intervention group will undergo a modified diagnostic pathway where a CAD-score ≤20 rules out stable CAD. If CAD-score >20 NIT is performed.
  Interventions: Device: CADScor®System

INTERVENTIONS:
Device: CADScor®System — The CADScor®System is a low cost, low resource-demanding, non-invasive, radiation-free device using highly advanced analysis of sounds originating from blood flow turbulence in the coronary circulation and myocardial motion. Heart sound recordings are obtained transcutaneously during a 3 minutes recording period with a microphone mounted at the IC4. A CAD-score on a scale from 0 to 99 is estimated immediately after the recording with a fully automated algorithm. The algorithm measures eight acoustic properties and the resulting acoustic score is combined with the clinical risk factors gender, age, and hypertension. The entire procedure lasts approximately 10 minutes.
  Arms: Intervention group

SUMMARY:
This study evaluates the addition of the CADScorSystem to a standard Diamond-Forrester score guided rule-out strategy in ambulatory patients referred with symptoms suggestive of stable coronary artery disease. Half of the patients will undergo stratification using a Diamond-Forrester score only, while the other half will undergo stratification using a Diamond-Forrester score and a CAD-score. The study hypothesis is that the addition of a CAD-score will reduce unnecessary testing without compromising patient safety.

DETAILED DESCRIPTION:
Purpose and Rationale for the Study:

The declining incidence of obstructive CAD and a good prognosis for patients with stable angina challenges the resource demanding approach recommended in current guidelines. The CADScor®System may be an efficient, fast and low-cost diagnostic tool with a high rule-out efficiency. The current study aims to investigate if the CADScor®System can be added as a rule-out test in patients referred with suspected stable CAD to reduce unnecessary testing

Study Hypothesis:

A Diamond-Forrester score plus CAD-score guided rule-out strategy is superior to a Diamond-Forrester score guided strategy alone in reducing diagnostic procedures and non-inferior in terms of safety outcomes in patients with symptoms suggestive of stable coronary artery disease.

Study Setting:

This study will enrol patients without known CAD who are referred with symptoms suggestive for stable CAD for outpatient evaluation at the participating sites. All patients will be symptomatic and require evaluation for suspected CAD. Thus, whether or not the patient chooses to participate in the study, the patient will undergo evaluation for suspected CAD. All the standard NIT modalities and ICA in the study are clinically well established and performed routinely and safely. Experimental testing involves the CADScor®System, for ruling out CAD before any NIT in the intervention group.

End of Study:

The study will end when all the following have occurred: (1) at least 2000 patients have been randomized, and (2) 12±1 months (1 year) have elapsed since the last patient was randomized.

Extended Follow-up after Study Termination:

Follow-up might be performed for up to 10 years after randomization. Follow-up information will be extracted from national registers, including information on cardiovascular events and treatments, hospitalizations and ambulatory visits due to cardiovascular events, and causes of death.

Statistical methods:

A detailed description of the planned statistical analyses will be documented in a separate statistical report and analysis plan (SAP), which will be completed before data base lock.

Sample size considerations:

A reduction of 15% or more in the primary endpoint is regarded as clinically significant. Assuming an alpha significance level of 0.05, a statistical power of 80% and an expected number of NIT/ICA of 0.94 per patient in the standard care group, a sample size of 314 patients in each arm is needed to ascertain superiority of the intervention.

A sample size of 1914 provides 90% power for testing non-inferiority in terms of MACE between the two testing strategies, at an alpha significance level of 0.05.

We choose to include 2000 patients, i.e. 1000 patients in each group, allowing for a 4% loss to follow-up and drop out and providing power for the primary endpoint and the secondary MACE non-inferiority endpoint.

Statistical analysis:

The full analysis set (FAS) will include all randomized patients in whom written informed consent was obtained and in accordance with the intention-to-treat principle all patients will be analysed according to the allocated treatment group.

The per-protocol set (PPS) will include only those patients from the FAS who did not have one of the following major protocol violations: inclusion criteria not met, exclusion criteria met, no DF-score calculation, or no CAD-score measurement (intervention group only). Patients who did not receive the randomly allocated CAD-score measurement will be included and analysed in the control group (per protocol analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Have signed the informed consent form.
2. Males and females, aged 30 years or above.
3. Be able and willing to comply with the clinical investigational plan.
4. Symptoms suggestive of stable coronary artery disease.
5. No history of coronary artery disease (prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft).

Exclusion Criteria:

1. Diamond-Forrester score >85%.
2. Prior non-invasive testing for stable CAD or invasive coronary angiography within 6 months of randomization.
3. Implanted donor heart, mechanical heart, mechanical heart pump.
4. Pacemaker or Cardioverter Defibrillator (ICD).
5. Implanted electronic equipment in the area above and around the heart.
6. Significant operation scars, abnormal body shape, fragile or compromised skin in the fourth left intercostal space recording area.
7. Receiving same day treatment with nitro-glycerine on the day of randomization.
8. Pregnancy.

The exclusion criteria '1. Diamond-Forrester score >85%' was removed after updating the study according to the 2019 ESC guidelines on chronic coronary syndrome. According to these current guidelines, no patients should be referred to invasive diagnostic test based on their PTP alone, and therefore is this exclusion criteria is no longer relevant.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2016 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Cumulative number of non-invasive and invasive diagnostic procedures | 1 year
  Difference between the two treatment groups in cumulative number of non-invasive and invasive diagnostic procedures. Non-invasive procedures include exercise electrocardiogram (ECG), cardiac computed tomography angiography (CCTA), Rubidium cardiac PET (Rb-PET), myocardial perfusion imaging (MPI), cardiac magnetic resonance imaging (CMRi) and stress echocardiography. Invasive procedures include invasive coronary angiography (ICA) only.

SECONDARY OUTCOMES:
Incidence of Major adverse cardiac events (MACE) | 1 year
  Difference between the two treatment groups in proportion of major adverse cardiac events. Major adverse cardiac events (MACE) are a composite of all-cause death, non-fatal myocardial infarction, unstable angina pectoris, heart failure, and ischaemic stroke.

OTHER OUTCOMES:
Change in chest pain | 3 months and 1 year
  Change in chest pain from baseline as assessed by the Seattle Angina Questionnaire (SAQ).
Change in quality of life | 3 months and 1 year
  Change in quality of life from baseline as assessed by the EuroQoL-5D.
First non-invasive tests | 1 year
  Difference between the two treatment groups in the number of first non-invasive testings.
Downstream tests | 1 year
  Difference between the two treatment groups in the number of downstream tests. Downstream tests are defined as all NITs and ICAs to detect CAD performed after a) DF-score and first standard non-invasive testing and b) DF-score, CAD-score and first non-invasive testing, respectively, in the two groups.
Invasive coronary angiographies (ICA) | 1 year
  Difference between the two treatment groups in the number of invasive coronary angiographies.
Negative invasive coronary angiographies | 1 year
  Difference between the two treatment groups in the number of negative invasive coronary angiographies.
Repeat referrals | 1 year
  Difference between the two treatment groups in the number of repeat referrals.
Time to rule-out CAD | 1 year
  Difference between the two treatment groups in time to rule-out CAD. Time to rule-out is assessed as the period from randomisation until the first test that rules out stable CAD.
Time to diagnosis of CAD | 1 year
  Difference between the two treatment groups in time to diagnosis of CAD. Time to diagnosis is assessed as the period from randomisation until the first test that leads to the final diagnosis.
Change in lifestyle measures | 3 months and 1 year
  Change in lifestyle measures from baseline as assessed by the HeartDiet questionnaire.
Optimal medical treatment | 1 year
  Difference between the two treatment groups in the proportion of patients initiating and adhering to optimal medical treatment (event prevention, antianginal therapy).
Incidence of individual components of MACE | 1 year
  Difference between the two treatment groups in the proportion of each of the individual components of major adverse cardiac events (all-cause death, myocardial infarction, unstable angina pectoris, heart failure, ischaemic stroke).
Cumulative contrast dose | 1 year
  Difference between the two treatment groups in the cumulative contrast dose.
Cumulative radiation dose | 1 year
  Difference between the two treatment groups in the cumulative radiation dose.
Bleedings requiring hospitalization | 1 year
  Difference between the two treatment groups in the proportion of bleedings requiring hospitalization.
Adverse events | 1 year
  Difference between the two treatment groups in the proportion adverse events related to the CADScor®System.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, DMSc., Principal Investigator — Bispebjerg og Frederiksberg Hospitaler; Søren Galatius, DMSc., Principal Investigator — Bispebjerg og Frederiksberg Hospitaler
Locations (6):
- Denmark (5):
  - Amager Hospital, Copenhagen S
  - University Hospital Herlev and Gentofte, Herlev
  - University Hospital Nordsjaelland, Hillerød
  - University Hospital Hvidovre, Hvidovre
  - University Hospital Bispebjerg and Frederiksberg, København NV
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bjerking LH, Hansen KW, Biering-Sorensen T, Bronnum-Schou J, Engblom H, Erlinge D, Haahr-Pedersen SA, Heitmann M, Hove JD, Jensen MT, Kruse M, Rader S, Strange S, Galatius S, Prescott EIB. Cost-effectiveness of adding a non-invasive acoustic rule-out test in the evaluation of patients with symptoms suggestive of coronary artery disease: rationale and design of the prospective, randomised, controlled, parallel-group multicenter FILTER-SCAD trial. BMJ Open. 2021 Aug 23;11(8):e049380. doi: 10.1136/bmjopen-2021-049380. PMID 34426466

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04121949/SAP_000.pdf